CLINICAL TRIAL: NCT01427361
Title: Prospective, Multi- Site, Clinical Study of Clinical Outcomes Following Hip Resurfacing Using VISIONAIRE Femoral Alignment Guide
Brief Title: Clinical Outcome of Birmingham Hip Resurfacing (BHR) Using VISIONAIRE Femoral Alignment Guide
Acronym: BHR
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: US-CR-135
Record Dates: First submitted 2010-08-06; First posted 2011-09-01 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to investigate the accuracy of the femoral implant placement utilizing the VISIONAIRE Femoral Alignment Guide in Birmingham Hip Resurfacing (BHR) surgery postoperatively after total hip resurfacing using the BHR System.

DETAILED DESCRIPTION:
This is a prospective, multi- site, clinical study of clinical outcomes following hip resurfacing using VISIONAIRE Femoral Alignment Guide. The objective of this study is to evaluate the safety and efficacy of the blocks and to assess alignment of the BHR system when using VISIONAIRE Femoral Alignment Guide. This study will also document any device-related surgical complications or adverse radiographic observations.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, at least 21 years of age, inclusive, and skeletally mature.
2. Patient diagnosed with osteoarthritis of the hip requiring primary total hip resurfacing due to:

   * Non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, traumatic arthritis, avascular necrosis, or dysplasia/DDH, or
   * Inflammatory arthritis such as rheumatoid arthritis.
3. Patient is willing to consent to participate in the study
4. Patient is in stable health and is free of or treated and stabilized for cardiac, pulmonary, hematological, or other conditions that would pose excessive operative risk.
5. Patient meets medical clearance to have surgery required for this study

Exclusion Criteria:

1. Patient with infection or sepsis.
2. Patient with any vascular insufficiency, muscular atrophy, or neuromuscular disease severe enough to compromise implant stability or postoperative recovery.
3. Patient is pregnant or plans to become pregnant during the course of the study.
4. Patient known to have insufficient bone stock to support the BHR device including:

   * Subjects with severe osteopenia should not receive a BHR procedure. Patients with a family history of severe osteoporosis or severe osteopenia.
   * Subjects with osteonecrosis or avascular necrosis (AVN) with >50% involvement of the femoral head (regardless of FICAT Grade) should not receive a BHR.
   * Subjects with multiple cysts of the femoral head (>1cm) should not receive a BHR.
   * Note: In cases of questionable bone stock, a DEXA scan may be necessary to assess inadequate bone stock.
5. Patient has known moderate to severe renal insufficiency. Subjects on medications (such as high-dose or chronic aminoglycoside treatment) or with co-morbidities (such as diabetes) that increase the risk of future, significant renal impairment should be advised of the possibility of increase in systemic metal ion concentration.
6. Patient has a known sensitivity to materials in the device.
7. Patient is immuno-suppressed.
8. Patient has physical, emotional or neurological conditions that would compromise the patient's compliance with postoperative rehabilitation and follow-up.
9. Patient has BMI >40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population considered for this study is patients requiring total hip resurfacing. The following inclusion and exclusion criteria will be used to identify study candidates.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Investigate the accuracy of the femoral implant placement utilizing the VISIONAIRE Femoral Alignment Guide in BHR surgery postoperatively after total hip resurfacing using the BHR System | 6 week
  Radiographic evaluation of postoperative femoral stem angle.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 week and 6 month
  Surgical and device related adverse events or revision

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - London Health Science Centers, London, Ontario
  - Sr. Michaels Hospital, Toronto, Ontario